CLINICAL TRIAL: NCT05274594
Title: Efficacy of Preoperative Radiotherapy for Non-responder Patients After Neoadjuvant Chemotherapy: a Pilot Observational Study
Brief Title: Efficacy of Preoperative Radiotherapy for Non-responder Patients After Neoadjuvant Chemotherapy
Status: Completed | Type: Observational
Sponsor: Istanbul Breast Society (Other)
Responsible Party: Sponsor
Other Study IDs: IstanbulBreast-22_01
Record Dates: First submitted 2022-01-30; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Breast Neoplasms; Radiotherapy; Complications; Survivorship; Breast Cancer
Keywords: breast neoplasm; radiotherapy; neoadjuvant therapy; chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy — Patients who are candidate for radiotherapy and received neoadjuvant chemotherapy for breast cancer were evaluated after neoadjuvant chemotherapy. Cases that do not have clinical response received radiotherapy before surgery in order to increase complete response.

SUMMARY:
Neoadjuvant chemotherapy (NACT) is widely used for locally advanced breast cancer cases. As the key factor is to achieve pathologic complete response (pCR), several physicians tried administering radiotherapy before surgery to increase response rates. In this single center observational cohort study, we aim to present the initial results as complete response rates and complication rates of additional neoadjuvant radiotherapy (NART) after NACT.

DETAILED DESCRIPTION:
Patients who received NACT were enrolled on the study depending on their order of admission. NACT regimen was 4 cycles of anthracycline and cyclophosphamide with 12 cycles of taxane based regimen. Trastuzumab for 12 monhts was also added if pathologically human epidermal growth factor receptor 2 (HER2+). This protocol was the same as planned for postoperative protocol and it was decided by the medical oncologist of the patient. Pathologic complete response (pCR) was defined as no residual invasive or in-situ tumor in the final pathology following neoadjuvant treatments. Clinical complete response (cCR) was defined as no sign of residual tumor mass and The Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria's were used to determine cCR. Patients were evaluated for clinical response between 4 and 6 weeks after the end of last NART. We waited as long as the NART period for clinical response evaluation of the cases.

Every patient was discussed in the preoperative multidisciplinary breast surgical oncology meeting before and after neoadjuvant treatment. The method of surgery was discussed in these meetings by a group of expert breast surgeons, plastic and reconstructive surgeons, radiation oncologists, medical oncologists, and radiologists. Patients were specifically evaluated for breast conservation, mastectomy or mastectomy with reconstruction. Likewise, the method of axillary surgery also discussed in these meetings. Indications for mastectomy were initially multi-centric tumors, large tumor volume relative to breast volume that is not allowing a good cosmetic result, patients with breast cancer related gene mutations, extensive in-situ component. Reconstruction with implant was also recommended to all mastectomy patients.

Radiotherapy was delivered via 4-6 megavoltage (MV) X-ray beam energies and Intensity Modulated Radiation Therapy (IMRT) or Volumetric Modulated Arc Therapy (VMAT) or forward planning IMRT (field in field - FinF) treatment techniques. NART was planned as 42.5 gray (Gy) in 16 fractions (with 10 Gy in 5 fractions sequential boost doses) or 50 Gy in 25 fractions (with 10 Gy in 5 fractions sequential boost doses) or 50.4 Gy in 28 fractions (with 59.9 Gy in 28 fractions simultaneous integrated boost doses) the whole breast irradiation plus nodal irradiation (including supraclavicular and axillary lymph nodes - Level I, II, III), if breast conserving surgery (BCS) is planned. If mastectomy is scheduled following NART, irradiation was planned with the same treatment volumes (the whole breast irradiation plus nodal irradiation) and doses like in BCS, but boost dose delivery was left to the radiation oncologist's preference. Radiotherapy to the mammary internal lymph nodes was delivered upon discretion of the radiation oncologist, and according to the tumor characteristics such as clinical stage or tumor location. Surgery was planned six weeks after the end of NART.

ELIGIBILITY:
Inclusion Criteria:

* American Joint Committee on Cancer (AJCC) clinical T1-3
* Biopsy proven N+
* Non-metastatic (M0)
* Patients who are planned to receive adjuvant radiotherapy at initial evaluation
* Patients who are candidate for neoadjuvant chemotherapy
* Patients who did not achieved clinical complete response after neoadjuvant chemotherapy

Exclusion Criteria:

* AJCC clinical T4
* AJCC Clinical N-
* AJCC Clinical M1
* Patients who achieved clinical complete response after neoadjuvant chemotherapy
* Patients who did not consent to have neoadjuvant radiotherapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients admitted to Istanbul Faculty of Medicine Breast Unit
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Complete response rate following neoadjuvant radiotherapy | Up to 4 weeks after definitive surgery
  Additional complete response effect of neoadjuvant radiotherapy for non-clinical complete responder patients following neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
Radiotherapy toxicity | During the first Four weeks after the last dose of radiotherapy
  Toxicity degree of neoadjuvant radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Müslümanoğlu, Prof. Dr., Principal Investigator — MD,FEBS,FACS
Locations (1):
- Istanbul Breast Society, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozkurt E, Sakai T, Wong SM, Tukenmez M, Golshan M. Survival Outcomes for Patients With Clinical Complete Response After Neoadjuvant Chemotherapy: Is Omitting Surgery an Option? Ann Surg Oncol. 2019 Oct;26(10):3260-3268. doi: 10.1245/s10434-019-07534-1. Epub 2019 Jul 24. PMID 31342356
- [Result] Bollet MA, Belin L, Reyal F, Campana F, Dendale R, Kirova YM, Thibault F, Dieras V, Sigal-Zafrani B, Fourquet A. Preoperative radio-chemotherapy in early breast cancer patients: long-term results of a phase II trial. Radiother Oncol. 2012 Jan;102(1):82-8. doi: 10.1016/j.radonc.2011.08.017. Epub 2011 Sep 8. PMID 21907436